CLINICAL TRIAL: NCT02535247
Title: A Phase I/II Study to Determine Feasibility and Safety MK-3475 Alone or in Combination With Copanlisib in Relapsed or Refractory NK and T-cell Non-Hodgkin Lymphoma
Brief Title: Study of MK-3475 Alone or in Combination With Copanlisib in Relapsed or Refractory NK and T-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Merck no longer providing drug for study
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-075
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — pembrolizumab; copanlisib

STUDY DESIGN:
Intervention Model Description: MK-3475 is given intravenously at a fixed dose of 200mg every 3 weeks. Copanlisib is given intravenously at RP2D determined from Phase I study 18 in cohort 1 (pembrolizumab alone; completed); 27 in Cohort 2; 4-12 in cohort 2a (phase I); 18 in cohort 2b (phase II). Total up to 48
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): MK-3475 given intravenously at a fixed dose of 200mg every 3 weeks for up to 36 cycles
  Interventions: Drug: MK-3475
- Combination (Active Comparator): MK-3475 is given intravenously at a fixed dose of 200mg every 3 weeks Copanlisib is given intravenously at RP2D determined from Phase I study
  Interventions: Drug: MK-3475; Drug: Copanlisib

INTERVENTIONS:
Drug: MK-3475
  Other Names: Pembrolizumab
Drug: Copanlisib
  Arms: Combination

SUMMARY:
This is a multicenter, single-arm, open label, study consisting of two cohorts. Cohort 2 explores the combination of copanlisib and pembrolizumab in patients with relapsed or refractory NKTCL, who have received at least 1 prior systemic therapy. Cohort 2 will include a phase 1 portion (cohort 2a) to determine the recommended phase 2 dose (RP2D) utilizing a standard 3+3 design, followed by a phase II portion where patients will be treated at the RP2D (cohort 2b). The primary endpoint for cohort 1 was progression-free survival; the primary endpoint for cohort 2a will be to determine RP2D for the combination therapy; and overall response rate at the end of 4 treatment cycles for cohort 2b. Patients will be assessed for response with PET CT or CT every 12 weeks using the revised Cheson criteria. Correlative endpoints will be exploratory and assess PD-1 expression on peripheral blood lymphocytes; peripheral blood T-cell and NK-cell functional assays; PD-1 and PD-L1 expression on tumor tissue; tumor infiltrating lymphocytes and gene expression panels using the nanostring technology as prognostic and predictive biomarkers, as well as monitoring of minimal residual disease via high-throughput sequencing of cell free tumor DNA, and exosome analysis.

DETAILED DESCRIPTION:
Patients with relapsed or refractory (RR) NK and T-cell Lymphoma (NKTCL), who have received at least 1 prior systemic therapy, were enrolled in cohort 1. The study design for cohort 1 was a single arm phase II 2-stage design, to explore monotherapy with the PD-1 antibody pembrolizumab (or MK-3475) given intravenously at a fixed dose of 200mg every 3 weeks for up to 36 cycles. Enrollment to this cohort has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed relapsed/refractory mature T-cell lymphoma that has progressed after a minimum of 1 systemic therapy with any of the following T-cell histologies:

   * Peripheral T-cell NHL, not other wise specified (PTCL, NOS)
   * Anaplastic large cell T-cell lymphoma (ALCL)
   * Anaplastic lymphoma kinase positive or negative
   * Angioimmunoblastic T-cell lymphoma
   * Subcutaneous panniculitis like T-cell lymphoma
   * Follicular T-cell lymphoma
   * Nodal peripheral T-cell lymphoma with TFH phenotype
   * Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL)
   * Enteropathy associated T-cell lymphoma
   * Hepatosplenic T-cell lymphoma
   * Extranodal NK/T-cell lymphoma, nasal type
   * Unclassifiable PTCL
   * Transformed cutaneous T-cell lymphoma (CTCL) to PTCL with systemic involvement (not local skin transformation).
2. Be willing and able to sign written informed consent for the trial.
3. Be at least 18 years of age on day of signing informed consent.
4. Have measurable disease based as defined by at least one lesion that can be measured in least 2 perpendicular dimensions and measures at least 1.5 cm in its long axis.
5. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion obtained within 28 days prior to study enrollment.
6. Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of treatment initiation.

   * Absolute neutrophil count (ANC) Greater than or equal to 1,500 /mcL, OR Greater than or equal to1,000 /mcL if lymphomatous bone marrow involvement Patients with documented marrow involvement may receive GCSF to achieve this value
   * Platelets greater than or equal to 100,000 / mcL, OR greater than or equal to 75,000 / mcL if lymphomatous bone marrow involvement Patients with documented marrow involvement may be transfused to this value.
   * Hemoglobin greater than or equal to 9 g/dL or greater than or equal to 5.6 mmol/L Patients with documented marrow involvement may be transfused to this value.
   * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) less than or equal to1.5 X upper limit of normal (ULN) OR greater than or equal to 40 mL/min for subject with creatinine levels greater than 1.5 X institutional ULN
   * Serum total bilirubin less than 1.5 X ULN OR Direct bilirubin less than the ULN for subjects with total bilirubin levels greater than 1.5 ULN
   * AST (SGOT) and ALT (SGPT) less than or equal to 2.5 X ULN OR less than or equal to 5 X ULN for subjects with liver involvement by lymphoma
   * Lipase less than or equal to 1.5 X ULN
   * International Normalized Ratio (INR) or Prothrombin Time (PT) less than or equal to 1.5 X ULN unless subject is receiving anticoagulant therapy
   * Activated Partial Thromboplastin Time (aPTT) less than or equal to 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.5.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of the first dose of treatment.
2. Patients diagnosed with Adult T-cell Leukemia/Lymphoma (ATLL) or T-cell PLL
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., worse than Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with worse than Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
7. Has known active intraparenchymal lymphomatous central nervous system (CNS) lesions and/or lymphomatous meningitis. Subjects with previously treated CNS involvement by lymphoma may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain lesions, and are not using steroids for at least 7 days prior to trial treatment.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjoegren's syndrome will not be excluded from the study.
9. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
18. Cohort 2a: Has received an allogeneic stem cell transplant. For cohort 2b, patients within the first 100 days of having undergone an allogeneic stem cell transplant will be excluded. Otherwise, patients who have received an allogeneic stem cell transplant are allowed as long as they have no evidence of active GVHD or are on immunosuppressive therapy
19. Uncontrolled arterial hypertension despite optimal medical management
20. Uncontrolled Type I or II diabetes mellitus as deemed appropriate by the investigator. Suggested guidelines for uncontrolled diabetes: HbA1c> 8.5%
21. Anti-arrhythmic therapy (beta blockers or digoxin are permitted)
22. Use of CYP3A4 inhibitors and inducers. Copanlisib is primarily metabolized by CYP3A4. Therefore concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from Day -14 of Cycle 1 until the Safety follow up visit. See Table in Appendix 5 for complete list
23. Concurrent diagnosis of pheochromocytoma
24. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
25. Prior exposure to PI3K inhibitors, unless on PI3K inhibitor therapy more than 6 months ago AND reason for discontinuation of prior PI3K inhibitor therapy was other than progression or toxicity.
26. Patients with detectable CMV viremia are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Fung, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Barta SK, Zain J, MacFarlane AW 4th, Smith SM, Ruan J, Fung HC, Tan CR, Yang Y, Alpaugh RK, Dulaimi E, Ross EA, Campbell KS, Khan N, Siddharta R, Fowler NH, Fisher RI, Oki Y. Phase II Study of the PD-1 Inhibitor Pembrolizumab for the Treatment of Relapsed or Refractory Mature T-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2019 Jun;19(6):356-364.e3. doi: 10.1016/j.clml.2019.03.022. Epub 2019 Apr 3. PMID 31029646

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: MK-3475 given intravenously at a fixed dose of 200mg every 3 weeks for up to 36 cycles
  MK-3475
- Combination: MK-3475 is given intravenously at a fixed dose of 200mg every 3 weeks Copanlisib is given intravenously at RP2D determined from Phase I study
  MK-3475
  Copanlisib
Period: Overall Study
Arm/Group | Treatment | Combination
Started | 17 | 0
Completed | 13 | 0
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Population: Study did not progress to portion with combination of pembrolizumab and copanlisib
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Combination | Total
Number analyzed (Participants) | 17 | 0 | 17
Age, Continuous [Median (Full Range); unit: years] | 71 [18 to 88] |  | 71 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 8 | 0 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Based on RECIST v1.1
Time Frame: 3 Months
Population: Some patients unevaluable for PFS
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 11 | 0
Participants | 6 |

2. Primary Outcome: Recommended Phase II Dose of the Combination of Pembrolizumab and Copanlisib
Time Frame: 6 months
Population: Study did not progress to portion with combination of pembrolizumab and copanlisib
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Determine Overall Response Rate by 4 Cycles of Combination of Pembrolizumab and Copanlisib
Time Frame: 6 months
Population: Study did not progress to portion with combination of pembrolizumab and copanlisib
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Time Frame: 6 Months
Population: Study did not progress to portion with combination of pembrolizumab and copanlisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 17 | 0
months | 3.2 [1.2 to 3.7] |

5. Secondary Outcome: Maximum Tolerated Dose of Pembrolizumab and Copanlisib
Description: Defined as the highest dose tested in which none or only one patient experienced dose-limiting toxicity (DLT) attributable to the study drug(s), when 6 patients have been treated at that dose and are evaluable for toxicity.
Time Frame: 6 months
Population: Maximum tolerated dose data not available because this data was not collected
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Expression of PD-1, PD-L1 and Tumor Infiltrating Lymphocytes (TIL) in Pre-treatment Tumor Specimens
Time Frame: 1 year
Population: Data was not collected as the trial was halted early after a preplanned interim futility analysis
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: PD-1 Expression and Leukocyte Activation Markers on Circulating Lymphocytes Pre-treatment
Description: PD-1 expression and leukocyte activation markers on circulating lymphocytes pre-treatment, at weeks 3 and 6, and at time of disease progression
Time Frame: Week 3
Population: Data was not collected as the trial was halted early after a preplanned interim futility analysis
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: PD-1 Expression and Leukocyte Activation Markers on Circulating Lymphocytes Pre-treatment
Description: as for outcome 7
Time Frame: Week 6
Population: Data was not collected as the trial was halted early after a preplanned interim futility analysis
Arm/Group | Treatment | Combination
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Study did not progress to portion with combination of pembrolizumab and copanlisib.
Arm/Group | Treatment | Combination
All-Cause Mortality (participants affected / at risk) | 11/17 | 0/0
Serious Adverse Events (participants affected / at risk) | 12/17 | 0/0
Other Adverse Events (participants affected / at risk) | 17/17 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=17) | Combination (N=0)
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Intractable vomiting (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Methicillin-Resistant Staphyloccus aureus infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Fever (General disorders) | 4 | 0
Sepsis (Infections and infestations) | 2 | 0
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Bilateral pneumonia (Infections and infestations) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Wound (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Neutropenic fever (Gastrointestinal disorders) | 1 | 0
Fecal impaction (Gastrointestinal disorders) | 1 | 0
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=17) | Combination (N=0)
Fatigue (General disorders) | 8 | 0
Fever (General disorders) | 8 | 0
Chills (General disorders) | 3 | 0
Edema limbs (General disorders) | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0
Injection site reaction (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Mucositis (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Abominal distension (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Oral hemmorhage (Gastrointestinal disorders) | 1 | 0
Generalized muscle eakness (Musculoskeletal and connective tissue disorders) | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 3 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Alkaline phosphatase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 2 | 0
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Blurred vision (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 2 | 0
Watering eyes (Eye disorders) | 2 | 0
Eye disorders - Other (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Vascular disorders - Other (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Congenital, familial and genetic disorders - Other (Congenital, familial and genetic disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT02535247/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT02535247/ICF_001.pdf